CLINICAL TRIAL: NCT00226629
Title: Evaluation of the Endovascular Repair for Aortic Aneurysm (EVAR) Program at LHSC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-03-155
Record Dates: First submitted 2005-09-23; First posted 2005-09-27 (Estimated); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Endovascular vs Open Repair

SUMMARY:
The purpose of this study is to compare the cost effectiveness, quality of life and outcomes of the endovascular stent graft repair with the open surgical repair of abdominal aortic aneurysms.

DETAILED DESCRIPTION:
Abdominal Aortic Aneurysms have been traditionally repaired using the standard open surgical technique. The use of Endovascular stent grafts(EVAR) to treat aortic aneurysms has been ongoing for approximately 8-10 years. Use of EVAR to treat aortic aneurysms in high risk has been reported to be beneficial. However, the costs of this therapy are quite significant and therefore in order to best understand the cost effectiveness of this type of aneurysm treatment, an extensive prospective comparative evaluation is required. This study will compare outcomes and cost-effectiveness for patients receiving EVAR, with high surgical risk, and OSR, with low surgical risk, and OSR, where there is high surgical risk and not suitable for EVAR based on anatomical complexity. Demographic, medical, health care resource utilization, cost, and quality of life information is collected from participating patients over a period of a year following repair.

ELIGIBILITY:
Inclusion Criteria:

* infrarenal abdominal aortic aneurysm,
* > 5.5 cm diameter
* scheduled for elective surgical repair

Exclusion Criteria:

* previous repair of AAA

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130
Dates: Start 2003-08 (Actual); Primary Completion 2006-06 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano DeRose, MD, FACS, FRCSC, Principal Investigator — LHSC, UWO